CLINICAL TRIAL: NCT05158257
Title: Clinical Of Plain Balloon Dilatation Combined Stent Versus Endovascular Debulking Combined Drug-coated Balloon to Treat Arteriosclerosis Occlusive Disease of Lower Extremity
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Xuanwu Hospital, Beijing (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: XuanwuH202110
Record Dates: First submitted 2021-10-07; First posted 2021-12-15 (Actual); Last update posted 2022-10-12 (Actual); Status verified 2022-10

CONDITIONS: Atherosclerosis; Ischemia
Keywords: stent; debulking; femoral artery; drug-coated balloon
MeSH Terms: conditions — Atherosclerosis; Ischemia | interventions — Stents

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention: balloon and Stents (Active Comparator): plain balloon and Stents group
  Interventions: Device: balloon and Stent
- Intervention: debulking and drug coated balloon (Experimental): debulking and drug coated balloon group
  Interventions: Device: endovascular debulking and DCB

INTERVENTIONS:
Device: balloon and Stent — balloon dilatation combined stent angioplasty
  Arms: Intervention: balloon and Stents
Device: endovascular debulking and DCB — endovascular debulking combined drug-coated balloon
  Arms: Intervention: debulking and drug coated balloon

SUMMARY:
This is a Prospective randomized controlled study to evaluate the difference of safety，effectiveness between endovascular debulking combined drug-coated balloon and balloon dilatation combined stent angioplasty in treatment of femoral-popliteal artery lesions.

DETAILED DESCRIPTION:
Prospective randomized controlled study to evaluate the difference of safety，effectiveness between endovascular debulking combined drug-coated balloon and balloon dilatation combined stent angioplasty in treatment of femoral-popliteal artery lesions. Patients with femoral-popliteal artery lesions in our department were randomly assigned to the endovascular debulking combined drug-coated balloon group and balloon dilatation combined with stent angioplasty group. Compare the ischemic improvement rate (limb salvage rate, postoperative patency rate) and the complications rate of two different treatments. At the same time, the peri-operative related factors that may affect the end point events, such as preoperative baseline data, lesion characteristics, imaging features, stent fracture, and end point observation indexes were analyzed by regression analysis.

ELIGIBILITY:
Inclusion criteria： 1.all patients signed an informed consent form; 2.digital subtraction angiography (DSA) revealed femoropopliteal artery stenosis above 70% or occlusion resulting in claudication (Rutherford clinical category-Becker class II-III2-3) or critical limb ischemia (CLI) (Rutherford clinical category 4-5-Becker class IV-V) 3.with unobstructed vascular inflow; 4.with at least a vessel runoff; 5. good compliance and regular follow-up.

Exclusion criteria: 1. Acute or subacute lower limb ischemia caused by acute intraluminal thrombus within the target lesion.; 2. Severe calcified lesions （grade 4 in the PACSS scale）; 3. In-stent restenosis lesion or surgical arterial bypass grafting; 4. Severe renal insufficiency: creatinine level greater than 2.5 mg/dL; 5. Platelet count below 100,000/μL or with antiplatelet / anticoagulation contraindications; 6. Immunologic diseases or malignant diseases; 7. Ongoing active infection; 8. Decompensated congestive heart failure or acute coronary syndrome; 9. Refuse to sign the informed consent Unwillingness to comply with follow-up suggestions.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 144 (Estimated)
Dates: Start 2021-09-30 (Actual); Primary Completion 2023-10-10 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
12-month Primary Patency Rate | 12 months
  systolic velocity ratio >2.4 as measured by Duplex ultrasound.

SECONDARY OUTCOMES:
Technical success rate | 1 day
  Technical success was defined as residual stenosis less than 30% by final
freedom from clinically-driven TLR rate | 12 months
  it is defined as the freedom from clinically-driven target lesion revascularization
Major Adverse Events at 12-month Post Procedure | 12 months
  Major adverse events included death, index limb ischemia, index limb amputation, clinically driven target lesion revascularization , and significant embolic events, which were defined as causing end-organ damage.
12-month Limb Salvage Rate | 12 months
  Limb Salvage is defined as the freedom from secondary major amputation

CONTACTS AND LOCATIONS:
Locations (1):
- Gu Yong Quan, Beijing, Beijing Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided